CLINICAL TRIAL: NCT05550454
Title: Comparison of Manual Ventilation and Automatic Mechanical Ventilation During Cardiopulmonary Resuscitation, Pilot & Feasibility Study
Brief Title: Cardiac Arrest and Ventilation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jong Hwan Shin, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAVE-I(P)
Record Dates: First submitted 2022-02-18; First posted 2022-09-22 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Advanced Cardiac Life Support; Ventilation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: It is a study conducted by random assignment to two groups of manual ventilation and automatic mechanical ventilation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Mechanical Ventilation (Experimental): Automatic Mechanical Ventilation during ACLS
  Interventions: Device: Automatic Mechanical Ventilation
- Manual Ventilation (Active Comparator): Standard care with manual ventilation, Ambu-bagging, during ACLS
  Interventions: Device: Manual Ventilation

INTERVENTIONS:
Device: Automatic Mechanical Ventilation — Ventilation settings:
  Mode: (S)Continuous Mandatory Ventilation Rate: 10 b/min. Tidal Volume: 500 ml (male), 450 ml (female) I:E=1:1 Positive end expiratory pressure (PEEP): 5 cmH2O Flow trigger: off Oxygen: 100% Alarms: Pressure 70 cmH20, Tidal volume 100 ~ 1,000 ml
  Arms: Automatic Mechanical Ventilation
Device: Manual Ventilation — Ambu-bagging (It is recommended in the guidelines as a ventilation method.) Methods: 10 times per minutes by medical personnel
  Arms: Manual Ventilation

SUMMARY:
Comparison of Manual Ventilation and Automatic Mechanical Ventilation during CPR, Pilot & Feasibility Study (CAVE-I trial)

DETAILED DESCRIPTION:
This is a preliminary randomized clinical trials comparing the effectiveness of the automatic mechanical ventilation method compared to manual ventilation methods commonly performed during advanced cardiac life support (ACLS) in emergency room for out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA)
* Transferred by only EMS without prehospital return of spontaneous circulation (ROSC)
* ACLS for at least 20 minutes in the emergency room
* Arterial blood gas analysis at least once during ACLS

Exclusion Criteria:

* In-hospital cardiac arrest (IHCA)
* Not transferred by Emergency Medical Service
* ROSC gained before arriving at the ER
* OHCA caused by trauma
* ACLS is not performed for more than 20 minutes because the death is obvious
* Not able to intubate the trachea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
ROSC: return of spontaneous circulation | Within 20 minutes of ACLS
  Rate of any ROSC after ACLS

SECONDARY OUTCOMES:
Arterial blood gas analysis (ABGA) parameters | The first test was conducted within 5 minutes of ACLS, and the second test 10 minutes after the first test.
  PH (no unit), PO2 in mmHg, PCO2 in mmHg, HCO3 in mEq/L
Ventilation parameters | During the entire ACLS time after randomization and endotracheal intubation
  Tidal volume (TV) and Minute volume (MV) during the entire ACLS

OTHER OUTCOMES:
Peak pressure (only in automatic mechanical ventilation group) | Randomized by automatic mechanical ventilation and during the entire ACLS time after endotracheal intubation
  Peak pressure of ventilator during the entire ACLS

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Metropolitan Goverment-Seoul National University Boramae Medical Center, Seoul, Korea (the Republic Of), South Korea

REFERENCES:
- [Derived] Shin J, Lee HJ, Jin KN, Shin JH, You KM, Lee SGW, Jung JH, Song KJ, Pak J, Park TY, Park CJ, Bae GT. Automatic Mechanical Ventilation vs Manual Bag Ventilation During CPR: A Pilot Randomized Controlled Trial. Chest. 2024 Aug;166(2):311-320. doi: 10.1016/j.chest.2024.02.020. Epub 2024 Feb 18. PMID 38373673